CLINICAL TRIAL: NCT04763291
Title: Effects of Long-term Consumption of Two Plant-based Dietary Supplements on Cardiovascular Health and Low-grade Inflammation in the Elderly
Brief Title: Cardiovascular and InflammAging Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Green Beat (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Lamprecht Manfred PhD, PhD, Principal Investigator, Green Beat
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 33-055 ex 20/21
Record Dates: First submitted 2021-02-02; First posted 2021-02-21 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Aging; Cardiovascular Diseases; Overweight or Obesity
Keywords: Aging; CVD prevention; Low-grade inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Overweight; Obesity | interventions — Vegetables

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group (No Intervention): Continue habitual diet and lifestyle.
- Fruit, Vegetable and Berry (FVB) group (Experimental): Participants have to ingest an encapsulated juice powder concentrate, otherwise continue their habitual diet and lifestyle.
  Interventions: Dietary Supplement: Juice Plus+ Fruit, Vegetable and Berry blends
- Omega group (Experimental): Participants have to ingest a plant-based fatty acid supplement, otherwise continue their habitual diet and lifestyle.
  Interventions: Dietary Supplement: Juice Plus+ Omega blend
- Fruit, Vegetable, Berry and Omega (FVBO) group (Experimental): Participants have to ingest an encapsulated juice powder concentrate along with a plant-based fatty acid supplement, otherwise continue their habitual diet and lifestyle.
  Interventions: Dietary Supplement: Juice Plus+ Fruit, Vegetable and Berry blends; Dietary Supplement: Juice Plus+ Omega blend

INTERVENTIONS:
Dietary Supplement: Juice Plus+ Fruit, Vegetable and Berry blends — Encapsulated juice powder concentrate derived from 36 dried fruits, vegetables and berries.
  Arms: Fruit, Vegetable and Berry (FVB) group; Fruit, Vegetable, Berry and Omega (FVBO) group
Dietary Supplement: Juice Plus+ Omega blend — Encapsulated plant-based fatty acid supplement.
  Arms: Fruit, Vegetable, Berry and Omega (FVBO) group; Omega group

SUMMARY:
Evidence from previous studies supports a strong relationship between fruit and vegetable consumption and reduced cardiac risk. This could be mediated via improvements on blood pressure, platelet function and vascular reactivity. Certain vitamins and polyphenols found in fruits and vegetables, have antioxidant and anti-inflammatory effects and play a major role on the function of immune cells. Previous studies have also demonstrated the importance of omega-3 fatty acids on humans' health and their positive effects on the cardiovascular system and blood lipids regulation, as well as their involvement on inflammatory response. Nutritional regimens with adequate intake of micronutrients, fruit and vegetables, omega-3 fatty acids, low in sugar and saturated fats, such as the Mediterranean diet or vegetarian diets, can reduce chronic inflammation and oxidative stress and improve cardiovascular risk profile. Considering that the population's fruit and vegetable and omega-3 intakes are below recommendations, whole food-based supplements could provide an accessible form of supplementation to bridge the gap between actual and recommended intakes. This study is aiming to assess whether long-term separate ingestions of an encapsulated juice powder concentrate and a plant-based omega fatty acid supplement, or a combined ingestion of the two, can affect biomarkers of cardiovascular health, low-grade inflammation and indicators of biological aging in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal
* Non-smokers
* BMI 18.5 to 40 kg/m2
* Vegetable intake ≤ 2 servings/ day
* Intake of fruits ≤ 2 servings /day
* Adherence to a 6-week washout period for dietary supplements not ingested for specific medical conditions.

Exclusion Criteria:

* Age <55 and >80 years
* Smokers (or ex-smokers who quit smoking less than 3 years ago)
* Aversion to stop the intake of multivitamins, multiminerals or omega fatty acid supplements
* Subjects with histamine intolerance
* Hypertension, starting with grade 2 according to the classification of the European Society of Hypertension: systolic blood pressure > 160mmHg, diastolic blood pressure >100 mmHg
* All medication taken for less than 3 months or with changes on the dosage over the last 3 months and medication for any of the conditions listed below.
* Clinically relevant infectious diseases
* Diabetes mellitus type I and type II
* Rheumatic diseases
* Auto-immune diseases
* Any stents and coronary artery diseases (CAD)
* Cancer patients
* Pregnancy
* Significant lifestyle changes, e.g. changes in diet or physical activity profile

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Lipid profile markers | 12 months
  Total cholesterol, HDL, LDL, ApoA1, triglycerides, Omega-3-Index
Hemostasis markers | 12 months
  Platelet aggregation, thrombelastometry, coagulation (Quick, PT, PTT)
Oxidative stress markers | 12 months
  oxLDL, MDA, carbonyl proteins, (CP), redox state of albumin, homocysteine
Glucose metabolism | 12 months
  Glucose, insulin, HOMA-IR, HbA1c
Concentration changes in cytokines/ cytokine receptors | 12 months
  TNF-α, sTNFR1 and sTNFR2, CCL5 = RANTES, IL-1β, hsCRP, CCL2 = MCP-1, Osteoprotegerin (OPG), IL-5, IL-8

SECONDARY OUTCOMES:
Vitamin K metabolism | 12 months
  Osteocalcin, matrix Gla protein (MGP), vitamins K1 and K2 (MK-7)
mitochondrial DNA copy number (mtDNA-CN) | 12 months
  mitochondrial DNA will be amplified and the ratio to genomic DNA will be calculated
Upper respiratory tract symptoms | 12 months
  The number of symptoms experienced and severity of symptoms will be assessed by the Wisconsin upper respiratory symptoms survey (WURSS).
Quality of life Questionnaire | 12 months
  Assessed through the Short Form Survey (SF-36), which consists of 8 scales, namely: physical functioning, physical role functioning, bodily pain, general health, vitality, social functioning, emotional role functioning, mental health. All items are scored on a scale from 0 to 100 and higher scores denote a more favourable health state.
Cognitive function | 12 months
  Cognitive function will be assessed by the CFD-index, which takes into account the following 5 dimensions: Attention (alertness, shared attention, processing speed), Verbal long-term memory, Executive functions (spatial working-memory, cognitive flexibility), Expressive language (word-fluency, object designation), Perceptual-motoric functions (visuoconstruction).
Neurotrophins | 12 months
  BDNF and NGF will be measured by ELISA

OTHER OUTCOMES:
Plasma concentrations of vitamins and carotenoids | 12 months
  Retinol, vitamins C, D, E (α-toc and γ-toc), α-carotene, β-carotene, lutein, zeaxanthin, lycopene, β-cryptoxanthin
Plasma concentrations of fatty acids | 12 months
  Docosahexaenoic acid, docosapentaenoic acid, eicosapentaenoic acid, arachidonic acid, alphalinolenic acid, linoleic acid, oleic acid, palmitoleic acid, stearic acid.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Lamprecht, PhD, Principal Investigator — Green Beat
Locations (2):
- Austria (2):
  - Green Beat, Graz
  - Otto Loewi Research Center, Section of Physiological Chemistry, Medical University of Graz, Graz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsiountsioura M, Cvirn G, Meixner-Goetz L, Ziegler T, Lamprecht M. Effects of long-term consumption of two plant-based dietary supplements on cardiovascular health and low-grade inflammation in middle-aged and elderly people: study protocol for a randomised, controlled trial. J Health Popul Nutr. 2023 Sep 19;42(1):100. doi: 10.1186/s41043-023-00434-x. PMID 37726820